CLINICAL TRIAL: NCT06225349
Title: Clinical Evaluation of the Improvement in Bioavailability of Four Magnesium-based Products in 40 Human Volunteers After an Oral Intake by Assessing Magnesium Absorption Kinetics in Plasma for 8 Hours
Brief Title: Clinical Evaluation of the Magnesium Absorption Kinetics in Human Plasma Upon Oral Intake of Magnesium-based Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionos Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MAGNESIUM_2023
Record Dates: First submitted 2024-01-17; First posted 2024-01-25 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers
Keywords: magnesium; plasma; bioavailability; oral; ingestion; ICP-MS; food; supplement
MeSH Terms: interventions — Dietary Supplements; Magnesium Oxide; magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Microencapsulated Magnesium (Experimental): This group will be provided with a the product Microencapsulated Magnesium.
  Interventions: Dietary Supplement: Dietary supplementation with Microencapsulated Magnesium
- Magnesium Oxide (Experimental): This group will be provided with a the product Magnesium Oxide.
  Interventions: Dietary Supplement: Dietary supplementation with Magnesium Oxide
- Magnesium Citrate (Experimental): This group will be provided with a the product Magnesium Citrate.
  Interventions: Dietary Supplement: Dietary supplementation with Magnesium Citrate
- Magnesium Bisglycinate (Experimental): This group will be provided with a the product Magnesium Bisglycinate.
  Interventions: Dietary Supplement: Dietary supplementation with Magnesium Bisglycinate

INTERVENTIONS:
Dietary Supplement: Dietary supplementation with Microencapsulated Magnesium — Volunteers will be provided with the product Microencapsulated Magnesium. For each volunteer, a blood sample from digital puncture will be obtained before (0 hour) and 1, 2, 4, 6, and 8 hours after oral intake of the product, and magnesium levels in plasma will be quantified by ICP-MS.
  Arms: Microencapsulated Magnesium
Dietary Supplement: Dietary supplementation with Magnesium Oxide — Volunteers will be provided with the product Magnesium Oxide. For each volunteer, a blood sample from digital puncture will be obtained before (0 hour) and 1, 2, 4, 6, and 8 hours after oral intake of the product, and magnesium levels in plasma will be quantified by ICP-MS.
  Arms: Magnesium Oxide
Dietary Supplement: Dietary supplementation with Magnesium Citrate — Volunteers will be provided with the product Magnesium Citrate. For each volunteer, a blood sample from digital puncture will be obtained before (0 hour) and 1, 2, 4, 6, and 8 hours after oral intake of the product, and magnesium levels in plasma will be quantified by ICP-MS.
  Arms: Magnesium Citrate
Dietary Supplement: Dietary supplementation with Magnesium Bisglycinate — Volunteers will be provided with the product Magnesium Bisglycinate. For each volunteer, a blood sample from digital puncture will be obtained before (0 hour) and 1, 2, 4, 6, and 8 hours after oral intake of the product, and magnesium levels in plasma will be quantified by ICP-MS.
  Arms: Magnesium Bisglycinate

SUMMARY:
The goal of this clinical trial is to study the effect of four magnesium-based products on the magnesium concentration in plasma of volunteers upon oral intake. 40 healthy volunteers will be on a low magnesium diet for 1 week; then, after a 8-hour fasting, a blood sample will be taken from a digital puncture before (0 hours) and 1, 2, 4, 6 and 8 hours after the oral intake of one of the products. This 1-week procedure (1 week diet, fasting, oral intake of the product and sample collection) will be repeated for all 4 tested products, summing a total of 4 weeks (1 week per product). On the day of the sample collection, volunteers will be provided with a standardized low-magnesium breakfast (1:15 hours after oral intake), low-magnesium lunch (6:15 hours after oral intake) and water ad libitum. All the meal plans (products, quantities and hours of the meals) will be identical in all the periods of the study. Plasma will be obtained from blood samples by centrifugation and the magnesium concentration in plasma will be measured by ICP-MS (inductively coupled plasma mass spectrometry).

DETAILED DESCRIPTION:
Magnesium is essential to the basic nucleic acid chemistry of all cells in all known living organisms. It is essential for DNA, RNA, and ATP synthesis, as well as for many other biological functions. Oral supplementation may improve the dietary intake of magnesium, which has been identified as a shortfall nutrient. In this study, the investigators will investigate the bioavailability of four magnesium-based products as food supplements by quantifying the magnesium levels in the plasma of volunteers after oral intake.

The study will be a double-blind trial to compare the bioavailability of four different magnesium products (Microencapsulated Magnesium, Magnesium Oxide, Magnesium Citrate and Magnesium Bisglycinate).

40 healthy volunteers between 20-55 years old will be enrolled in the study. Volunteers will be on a low magnesium diet for 1 week, including the consumption of low mineralization water; then, after a 8-hour fasting, a blood sample will be taken from a digital puncture before (0 hours) and 1, 2, 4, 6 and 8 hours after the oral intake of one of the products. This 1-week procedure (1 week diet, fasting, oral intake of the product and sample collection) will be repeated for all 4 tested products, summing a total of 4 weeks (1 week per product). On the day of the sample collection, volunteers will be provided with a standardized low-magnesium breakfast (1:15 hours after oral intake), low-magnesium lunch (6:15 hours after oral intake) and water ad libitum. All the meal plans (products, quantities and hours of the meals) will be identical in all the periods of the study. After every sample collection, participants will be allowed to leave the clinic, and asked to return at the required time-points. Volunteers will be requested not to practice any sport or to take part in any kind of strenuous exercise/activity during the day of collection.

Blood samples will be taken by digital puncture (non-invasive fingerstick procedure, by using VeriFine safety lancets 21G). The blood samples will be collected in EDTA-containing tubes (Minicollect tube K3E EDTA), centrifuged at 1000 rpm, 5 minutes at 4ºC, and plasma (supernatant) will be collected. Then, the magnesium levels in plasma will be measured by mass spectrometry ICP-MS (Mass Spectrometry with Inductively coupled plasma). The plasma samples of the 8-hour time point will not be analyzed by ICP-MS in principle, instead the samples will be stored at -80ºC and may be analyzed in further stages of the project.

There will be no consumption of supplements or specific food containing high levels of magnesium in the previous 7 days before the beginning of the experiment and during the experiment. Low mineralization water will be provided to the volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 20 and 55 years of all races/ethnicities.
* Body mass index of 18-35 kg/m2.
* Last participation in a clinical study of this type must be at least 15 days before the start of this study.
* Fasting conditions during 8 hours before the experiment (with the exception of low mineralization water).
* No consumption of food supplements or specific food containing high levels of magnesium (see attachment) during the week before the start of the treatment.

Exclusion Criteria:

* People with gastrointestinal diseases (diabetes, gastritis, Crohn's disease, celiac disease, ulcers, intolerances, etc.).
* People with cardiorespiratory diseases (chronic bronchitis, chronic obstructive pulmonary disease, pulmonary emphysema, asthma and bronchiectasis, thrombi, heart disease, heart disorders, arrhythmias, insufficiencies, etc.).
* Pregnant or lactating women or who plan to become pregnant during the study.
* People under medical treatment in the weeks prior to the study that could interfere with the evaluations of the present study (according to the investigator's criteria).
* People who are within a dietary period outside their usual habit.
* People who demonstrate manifest incapacity to understand or follow the protocol or the informed consent.
* Allergy or reactivity to any of the components of the product, or to a product with a category similar to the tested one.
* Surgically operated for a heart condition.
* People with forecast of changing routine or relevant way of life, during the period of the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-28 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Quantification of the changes of the magnesium levels in plasma of volunteers at time 0 hours (before consuming the product), and 1, 2, 4, 6, and 8 hours after oral intake of the product. | Upon oral intake, blood samples will be obtained by digital puncture at each time point; time 0 hours (before consuming the product), and 1, 2, 4, 6, and 8 hours after oral intake of the product.
  40 healthy volunteers will be on a low magnesium diet for 1 week; then, after a 8-h fasting, a blood sample will be taken from a digital puncture before (0 hour) and 1, 2, 4, 6 and 8 hours after the oral intake of one of the products. This 1-week procedure (1 week diet, fasting, oral intake of the product and sample collection) will be repeated for all 4 tested products, summing a total of 4 weeks (1 week per product). Blood samples will be taken by digital puncture (non-invasive fingerstick procedure, by using VeriFine safety lancets 21G). The blood samples will be collected in EDTA-containing tubes (Minicollect tube K3E EDTA), centrifuged at 1000 rpm, 5 minutes at 4ºC, and plasma (supernatant) will be collected. Then, the magnesium levels in plasma will be measured by mass spectrometry ICP-MS (Mass Spectrometry with Inductively coupled plasma) and expressed in mg magnesium per liter.

CONTACTS AND LOCATIONS:
Overall Officials: David Pajuelo Gamez, PhD, Principal Investigator — Bionos Biotech S.L.
Locations (1):
- Bionos Biotech S.L., Valencia, Spain

IPD SHARING:
Plan to Share IPD: No